CLINICAL TRIAL: NCT04801121
Title: Fetal Growth and Placental Function in Pregnancies Complicated by Diabetes
Acronym: FaPDi
Status: Unknown | Type: Observational
Last Known Status: Enrolling by invitation
Sponsor: Sidsel Linneberg Rathcke (Other)
Collaborators: Aarhus University Hospital (Other); University of Nottingham (Other)
Responsible Party: Sponsor-Investigator, Sidsel Linneberg Rathcke, MD, PhD student, Aalborg University Hospital
Organization: Aalborg University Hospital (Other)
Other Study IDs: N-20200065
Record Dates: First submitted 2021-03-08; First posted 2021-03-16 (Actual); Last update posted 2022-07-26 (Actual); Status verified 2022-07

CONDITIONS: Pregnancy in Diabetics; Placenta; Fetal Growth; Magnetic Resonance Imaging
Keywords: Pregestational diabetes; Placenta dysfunction; Placenta pathology; Abnormal fetal growth; Functional magnetic resonance imaging; 3D volume magnetic resonance imaging
MeSH Terms: conditions — Pregnancy in Diabetics

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 9 Months
Biospecimen Retention: Samples With DNA — Blood samples from participant, Umbilical cord blood samples, Placental tissues biopsies
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Pregestational diabetic pregnant: Cases: Women with type 1 or type 2 diabetes before start of pregnancy
- Non-diabetic pregnant: Controls: Women without metabolic disease before start of pregnancy

SUMMARY:
Diabetic pregnancies are often complicated by placental dysfunction with reduced transfer of oxygen from the mother to the fetus, which may compromise fetal growth and organ development. In diabetic pregnancies, hyperinsulinemia and hyperglycemia very often leads to fetal macrosomia. The combination of reduced placental oxygen transfer and increasing fetal demand due to fetal overgrowth may possess a particular risk of adverse pregnancy outcome.

Current methods in the antenatal identification of placental dysfunction relies on estimates of fetal size and fetal wellbeing using ultrasound including Doppler flows measurements. These measurements are only indirect estimates of placental function, as no clinical method exists to assess placental function directly. In diabetic pregnancies, the estimates are further limited due to fetal overgrowth and unreliable Doppler. In addition, in diabetic pregnancies, intrauterine fetal weight estimates by ultrasound are inaccurate because of asymmetric fetal growth. Therefore, new accurate methods to assess placental function, fetal oxygenation and fetal growth in this particular group of high-risk pregnancies is highly needed. Early and precise identification of pathology in diabetes pregnancy may lead to an improved outcome in the offspring, as precise identification of pathology facilitates important obstetric decisions in regards to maternal antidiabetic treatment and timing of delivery. Resent research indicates that MRI is useful for this purpose.

It is well described, that preeclampsia is associated with an increased maternal risk of cardiovascular disease later in life. Recent studies suggest, that pregestational subclinical cardiovascular dysfunction, in particular left ventricular dysfunction, may increase the risk of preeclampsia and fetal growth restriction during pregnancy. Cardiac MRI is a sensitive method to detect subclinical maternal cardiac dysfunction, which may be used in identification of high-risk pregnancies. In addition, the longitudinal design of this study allows for the investigation of cardiovascular changes during pregnancies in normal pregnancies and pregnancies complicated by diabetes.

The overall aim of this study is to improve the antenatal fetal and maternal monitoring in diabetes pregnancies. Early and precise identification of pregnancy pathology provides a better basis for important obstetric decisions regarding antidiabetic treatment, monitoring intervals and timing of delivery, which leads to a better outcome for the mother and offspring.

Hypothesis

Project A:

Placental function and fetal oxygenation in diabetic pregnancies estimated by T2* weighted placental and fetal MRI

Aim: To investigate placental function and fetal oxygenation by longitudinal T2* weighted placental MRI and the association with pregnancy complications.

Hypothesis:

* Diabetic pregnancies are characterized by placental hypoxia (low T2* value)
* Diabetic pregnancies are characterized by fetal hypoxia (low T2* value)
* Fetal and placental hypoxia is a risk factor of placental related complications in pregnancy such as low birth weight, preterm delivery, acute cesarean sections and preeclampsia.

Project B: Fetal growth and the growth of selected fetal organs in diabetic pregnancies estimated by longitudinal MRI volumetry

Aim: To investigate growth velocity of the fetus and selected fetal organs and the correlation with pregnancy complications.

Hypothesis:

* Diabetic pregnancies are characterized by accelerated fetal growth in the third trimester
* Diabetic pregnancies are characterized by asymmetric growth (reduced brain/liver-volume ratio)
* Abnormal fetal growth is associated with dysregulated maternal diabetes.
* Abnormal fetal growth is a risk factor of pregnancy complications such as; macrosomia, preterm delivery and acute cesarean sections.

Project C:

Maternal cardiac function in diabetic pregnancies estimated by MRI

Aim: To investigate maternal cardiac function and the correlation with pregnancy complications such as preeclampsia and fetal growth restriction.

Hypothesis:

* Maternal cardiac function is altered in diabetes pregnancies when compared to normal pregnancies.
* Impaired cardiac function (left ventricular dysfunction) is a risk factor of preeclampsia and fetal growth restriction.

DETAILED DESCRIPTION:
Maternal diabetes is an increasing problem among pregnant women worldwide. The incidence of diabetes in pregnancy has increased by 50% during the last 20 years, which is related to increased maternal BMI and higher maternal age. In Denmark the current incidence of gestational diabetes is approximately 6%. Maternal diabetes is a serious complication of pregnancy, and it is associated with an increased risk of maternal and neonatal complications such as preeclampsia, abnormal fetal growth, fetal asphyxia, still birth, caesarian section and premature delivery. In addition, diabetes is associated adverse long term consequences in the mother and the offspring such as increased risk of diabetes and cardiovascular disease.

These complications may be related to impaired fetal oxygenation, which is a result of increased oxygen demand of the macrosomic fetus and impaired fetal supply of oxygen due to placental dysfunction. The diabetic placenta is characterized by immaturity and maternal vascular malperfusion which leads to a reduced transport of oxygen from the mother to the fetus. At the same time, there are adaptive changes such as peripheral vascular hyperplasia, which tends to normalize the oxygen transport capacity. However, in a number of diabetic pregnancies this process remains inadequate to meet the increasing metabolic demand of the growing fetus. This explains why diabetic pregnancies have an increased risk of chronic intrauterine hypoxia and asphyxia in labor.

Current antenatal care in pregnancies complicated by diabetes focus on keeping maternal glucose level stable by the use of either diet or insulin treatment. It has been demonstrated that maternal glucose control is directly related to placental development and adverse obstetric outcomes. Placental function or fetal oxygenation cannot be assessed directly by current clinical methods. In antenatal care screening for placental dysfunction focus on ultrasound estimates of fetal size and ultrasound Doppler measurement of fetal and umbilical blood flow. Small fetal size and specific circulatory changes are indirect signs of placental dysfunction. Unfortunately, in diabetic pregnancies, screening for placental dysfunction is limited by fetal macrosomia and unreliable Doppler flow measurements and therefore new methods to directly assess placental function and fetal growth in this particular group of high risk pregnancies is highly needed in order to ensure rational obstetric decisions on when and how to deliver these high-risk fetuses.

It is well described, that preeclampsia is associated with an increased maternal risk of cardiovascular disease later in life. Women with GDM has a substantially increased risk of both preeclampsia and cardiovascular disease and GDM may be recognized as an early marker of atherosclerosis . Recent studies suggest, that pregestational subclinical cardiovascular dysfunction, in particular left ventricular dysfunction, may increase the risk of preeclampsia and fetal growth restriction during pregnancy. Therefore, early identification of maternal cardiovascular dysfunction is highly important, as prophylactic treatment with aspirin before gestational week 16 may reduce the risk of preeclampsia by more than 50%. Cardiac MRI is a sensitive method to detect subclinical maternal cardiac dysfunction, which may be used in identification of high-risk pregnancies. In addition, the longitudinal design of this study allows for the investigation of cardiovascular changes during pregnancies in normal pregnancies and pregnancies complicated by diabetes.

The overall aim of this study is to improve the antenatal fetal and maternal monitoring in diabetes pregnancies. Early and precise identification of pregnancy pathology provides a better basis for important obstetric decisions regarding antidiabetic treatment, monitoring intervals and timing of delivery, which leads to a better outcome for the mother and offspring.

Hypothesis

Project A:

Placental function and fetal oxygenation in diabetic pregnancies estimated by T2* weighted placental and fetal MRI

Aim: To investigate placental function and fetal oxygenation by longitudinal T2* weighted placental MRI and the association with pregnancy complications.

Hypothesis:

* Diabetic pregnancies are characterized by placental hypoxia (low T2* value)
* Diabetic pregnancies are characterized by fetal hypoxia (low T2* value)
* Fetal and placental hypoxia is a risk factor of placental related complications in pregnancy such as low birth weight, preterm delivery, acute cesarean sections and preeclampsia.

Project B: Fetal growth and the growth of selected fetal organs in diabetic pregnancies estimated by longitudinal MRI volumetry

Aim: To investigate growth velocity of the fetus and selected fetal organs and the correlation with pregnancy complications.

Hypothesis:

* Diabetic pregnancies are characterized by accelerated fetal growth in the third trimester
* Diabetic pregnancies are characterized by asymmetric growth (reduced brain/liver-volume ratio)
* Abnormal fetal growth is associated with dysregulated maternal diabetes.
* Abnormal fetal growth is a risk factor of pregnancy complications such as; macrosomia, preterm delivery and acute cesarean sections.

Project C:

Maternal cardiac function in diabetic pregnancies estimated by MRI

Aim: To investigate maternal cardiac function and the correlation with pregnancy complications such as preeclampsia and fetal growth restriction.

Hypothesis:

* Maternal cardiac function is altered in diabetes pregnancies when compared to normal pregnancies.
* Impaired cardiac function (left ventricular dysfunction) is a risk factor of preeclampsia and fetal growth restriction.

Predictors in general

Project A:

Placental function and fetal oxygenation in diabetic pregnancies estimated by T2* weighted MRI

The following predictors will be compared between the study groups:

Predictors:

* T2* values in the placenta, as a marker for placental hypoxia
* T2* values in the fetus, as a marker for fetal hypoxia
* Maternal serum markers of placental dysfunction
* Maternal glucose regulation (HgbA1c)

Project B:

Fetal growth and the growth of selected fetal organs in diabetic pregnancies estimated by longitudinal MRI volumetry

The following predictors will be compared between the study groups:

Predictors:

* Total volume of the fetus (MRI volumetry)
* Total volume of the brain and liver, as well as brain/live-volume ratio (MRI volumetry)
* Maternal glucose regulation (HgbA1c)

Project C:

Maternal cardiac function in diabetic pregnancies estimated by MRI

The following predictors will be compared between the study groups:

Predictors:

* Maternal cardiac function (Cardiac MRI)
* Maternal glucose regulation (HgbA1c)
* Maternal serum markers of placental and cardiac dysfunction

Method

Study design: Clinical prospective study Inclusion period: October 1st 2020 - September 30th 2023 Place: Department of Obstetrics and Gynecology, Aalborg University Hospital (AaUH) The longitudinal design of this study allows formation of trajectories of T2* values and fetal growth in normal pregnancies as well as subtypes of diabetes pregnancies.

Patient inclusion and exclusion:

The following groups are included at the Department of Obstetrics and Gynecology, AaUH

1. Pregestational diabetes (PGDM) (n=50)
2. Uncomplicated pregnancies (UP) (n=50)

   Inclusion criteria:
   * Age >18 years
   * Singleton pregnancy

   Exclusion criteria:
   * Fetal malformation or abnormal karyotype
   * Maternal height from spine to chest > 43 cm (for technical reasons)
   * Sever claustrophobia or any other contradictions to MRI
   * Women who do not read or understand Danish

   Recruitment and informed consent:

   All pregestational diabetes and uncomplicated pregnancies who meet the above-mentioned inclusion criteria will be presented for the project by the obstetrician/sonographer performing the ultrasound at their first trimester scan. It will be emphasized that participating is optional, rejection of participating will not affect the ongoing or future treatment of the women and the women can withdraw their consent at any time without reason. The results of the project examination are for research only, and they will not affect the clinical decisions regarding the current pregnancy.

   If interested the woman will receive written information. The written information consists of the document "Written participant information" and "Subjects' rights in a health science research project". She will then have time to read and consider the information carefully. If the woman is still interested in participating in the project, she will receive oral information about the project and about her rights as a trial subject by the doctor responsible for the project (PhD student Sidsel Linneberg Rathcke). The woman has the right to have another person with her during the oral information. The oral information will be given when the woman is ready for additional information. The oral information will be given in one of the departments outpatient rooms, where the information can be given undisturbed and in private. The oral information can be given at the same day as the written information or another day depending on the woman. The woman will have at least 24 hours of consideration prior to giving informed consent. The written consent will give the research team access to the patient's chart and all the information's regarding the patient's health necessary to complete, monitor and control the project. The woman can retract the informed consent at any time and without a reason, and this will not affect the following examinations or treatment during the pregnancy. Moreover, participation will not prevent or postpone necessary treatment and all participants will still attend in their regular pregnancy controls both in and out of the department / hospital.

   Participants will have to give an additional informed consent to give the permission to store the remaining blood, a blood sample from the umbilical cord and a small section of the placenta tissue in a clinical biobank for future research projects. This consent can be retracted at any time and the blood/placenta tissue will then be disposed. This decision is independent of the participation in the rest of the project described in this protocol.

   Study outline:

   All women will have three antenatal examinations and one postnatal examination. The examinations are outlined below and described in the following.

   Antenatal examination GA 14-16, 26-30 and 35-38
   * MRI examination: Fetal, placental and maternal cardiac scan.
   * Ultrasound: Fetal weight estimate and Doppler flow measurements of uterine, fetal and umbilical blood flow
   * Maternal blood sample - serum markers and electrocardiogram (ECG)

   Postnatal examination
   * Clinical information: Obstetric interventions, maternal and fetal outcomes, birth weight
   * Cord blood sample - serum markers
   * Maternal blood sample - serum markers
   * Histopathological placental examination

   MRI The MRI scan will be performed at Aalborg University Hospital North. The scan is performed with the pregnant woman in a left lateral position and she must wear hearing protection during the scan. The MRI examination time is 30 - 45 minutes. Any potential influence on the fetus are explained in the section MRI safety.

   The MRI scan includes the following assessments:
   * T2* weighted MRI of the placenta and the fetus
   * Volumetry of the placenta, the total fetus and selected fetal organs such as the fetal brain and liver.
   * Maternal cardiac MRI
   * Left ventricle end-diastolic volume index
   * Right ventricle end-diastolic volume index
   * Left ventricle end-systolic volume index
   * Right ventricle end-systolic volume index
   * Left ventricle ejection fraction (EF)
   * Right ventricle ejection fraction (EF)
   * Cardiac output (CO)
   * Left ventricle mass index, end-diastolic diameter and wall thickness
   * Native T1 mapping of the myocardium
   * Systolic myocardial deformation: longitudinal, circumferential, and radial

   Ultrasound The ultrasound examination will be performed at Aalborg University Hospital North. The ultrasound examination time is 30 minutes. The ultrasound scan will include Doppler flow assessments of the uterine artery (UtA), umbilical artery (UA) and the middle cerebral artery (MCA) and an ultrasound estimate of the fetal weight by fetal biometrics using Hadlock formula.

   Maternal serum markers and ECG A venous blood sample will be collected from the woman on the day of MRI and at the day of birth. The blood sample will be analyzed immediately for maternal baseline physiology (glucose, HgbA1c, electrolytes, liver parameters, hematological parameters), and will be used to compare blood glucose regulation between the groups. At the end of the inclusion period, all blood samples will be analyzed for specific placental and cardiac markers. The blood samples will be stored at Department of Clinical Biochemistry, Aalborg University Hospital until analysis.

   The remaining blood will be stored in a biobank for future research if the woman gives her permission.

   An ECG will be obtained from the woman on the day of MRI.

   Clinical information Maternal and pregnancy characteristics as well as pregnancy outcomes are collected from the clinical record.

   Maternal characteristics
   * BMI, age, ethnicity
   * Smoking status
   * Mode of conception
   * Parity

   Current pregnancy
   * Fetal
   * Growth
   * Malformation and chromosomal abnormalities
   * Maternal
   * Blood pressure
   * Urine samples
   * Blood sugar profile
   * Glucose regulation (HgbA1c)
   * Medication - anti-diabetes treatment (diet, insulin dose)
   * Serum markers from nuchal scan: PAPP-A and hCG
   * Gestational diabetes (OGGT level at 2 hours)
   * Pregnancy complications

   Delivery
   * Gestational age at birth
   * Induction of labour
   * Instrumentation, cesarean section (acute/elective)
   * Mode of delivery
   * Neonatal
   * Status (live/dead)
   * Admission to Neonatal Intensive Care Unit (days)
   * Apgar score
   * Umbilical cord pH
   * Sex
   * Birth weight, length, head and abdominal circumference
   * 2-hour blood glucose
   * Placenta
   * Weight, pathology report

   Umbilical cord blood serum markers A blood sample from the umbilical cord will be collected when the routine blood samples for pH-analysis are taken. This additional blood sample will be stored in a biobank for future research, regarding fetal glucose metabolism, fetal growth and placental function, if the woman gives her permission.

   Placental histopathological examination A trained pathologist will examine all the placentas postnatally. The examination will be done according to the national standard protocol. The pathologic examination of the placenta includes macroscopic and microscopic evaluation for signs of maternal and/or fetal malperfusion which indicates placental dysfunction. The pathologist will be blinded to clinical information- except gestational age at birth A placental biopsy will be stored in a biobank for future research if the woman gives her permission.

   Power calculation Due to lack of presumptions for power calculations, the number of women to be included in this study is based on the estimated number of women available and the clinical relevance.

   AaUH is a tertiary center for diabetes in pregnancy. The total number of deliveries is 3700 pr. year, and the number of pregnancies complicated by pregestational diabetes every year is around 60. Previous clinical studies on Placental MRI conducted at AaUH have demonstrated an inclusion success ratio of 70%. Thus, it should be feasible to include the estimated number of participants during the 2-year recruitment period.

   Ethics and risks

   Data handling Personal data are anonymized by an encrypted ID-number and data is stored in at Aalborg University Hospital in a locked cabinet in a locked room on a device locked by a code. An MRI database is established in RedCap.

   Data collection is approved by a regional notification to The Danish Data Protection Agency. All data will be handled in compliance with the General Data Protection Regulation (GDPR) and the Data Protection Act.

   MRI safety MRI is a widely used method to examine the fetus if any structural malformation (e.g. cerebral) or invasive placental disorders is suspected during ultrasound examination. Then an MRI with 1.5 Tesla magnetic field are performed to give additional information to the ultrasound previously done. Present data have not documented any harmful effects of MRI during pregnancy and no studies have shown any association between MRI and adverse fetal outcome. The potential harmful effects are discussed below.
   * Acoustic noise The MRI scanner generates noise in the range from 80 to 120 dB during acquisition of images. Ear protection is recommended for adults at this level of noise. The fetus is protected by the maternal abdomen and by the amniotic fluid, which reduces fetal noise exposure with at least 30 dB . The Danish Working Environment Authority suggests that 85 dB during a workday for pregnant women is likely to affect the fetus. No studies have shown hearing impairment of fetuses exposed to 1.5 T MRI during pregnancy.
   * Radiation and static magnetic fields MRI does not involve ionizing radiation. Static magnetic fields may interact with living tissues in various ways with one important mechanism being the magnetic induction, which may create electric currents by moving electrolytes in the blood vessels. No change in heart rate or systolic/diastolic blood pressure have been demonstrated when humans were exposed to 8 T for 1 hour. Likewise, studies using cardiotocography have demonstrated no effects on fetal heart rate during MRI. Another mechanism is the magneto-mechanical effect from static magnetic field, which induces reorientation of molecules. However, the magneto-mechanical effect is considered too small to affect human tissue in vivo, since human tissue does not contain strong ferromagnetic components. According to a review by the International Commission on Non-Ionizing Radiation Protection (ICNRIP), no consistent effects of static magnetic field exposure on reproduction and development have been seen in mammalian species.
   * Tissue heat The radiofrequency pulses used for generating the MR images may deposit heat in the tissues. Therefore, during the MRI acquisition a specific absorption rate (SAR value, Watt/kg) is calculated in order to prevent tissue heating. The SAR value will estimate the amount of thermal energy conducted and correlates to the tissue heat deposited. The SAR value is directly correlated to the time of the MRI scan. According to the recommendations by the International Commission on Non-Ionizing Radiation Protection (ICNIRP) , the whole-body SAR value should be kept below 2 W/kg during a one hour scan equivalent to a raise in adult tissue temperature of 0.5°C and a rise of fetal temperature to less than 38°C. Within a 1.5 T MRI system, the fetal peak SAR value is approximately 50% of that generated in the mother and using standard sequences at 1.5 T for less than one hour, the SAR value does not exceed the recommended maximum value, neither for the mother nor the fetus.

   Ultrasound safety Thermal effects of ultrasound examination have been investigated and a temperature elevation of 1.5°C is generally considered as the threshold and safe for the fetus .

   Thermal Index (TI) is the prediction of the temperature rise in the tissue within the ultrasound beam. TI is depending on ultrasound frequency, focus of the beam and duration of exposure. Perfusion, absorption and reflection of the tissue affect the temperature of the tissue. TI is a relative risk for the temperature rise and is expressed TI = 1.0 if the ultrasound beam may cause a temperature rise of 1°C. A rise of more than 1°C in the tissue may cause biological effects42. TI remains very low and under 1.0 during routine obstetric ultrasound examinations .

   No adverse effects in humans have been showed when exposed to diagnostic ultrasound.

   Research ethical considerations None of the examinations during this project will cause harmful effect neither for the pregnant woman or the fetus. The woman should attend the regular antenatal care program. None of the examinations during this project will affect or delay the clinical decisions.

   Longitudinal T2* weighted placental and fetal MRI, volumentry MRI and maternal cardiac MRI are all methods that need to be validated in diabetes pregnancies. Therefore, the MRI data analysis is blinded to clinical information, and the MRI will not contribute to any clinical decisions during the current pregnancy. However, the knowledge obtained by this study may improve the general antenatal care in a longer perspective.

   Clinical perspectives Pregnant women with diabetes possess a group in particular high risk of placental related complications of pregnancy. MRI may improve the antenatal care as the current methods based on ultrasound measurements of fetal growth and fetal circulation are inadequate. MRI provides precise estimates of fetal oxygenation, placental function and maternal cardiac function to support the obstetric decisions.

   Early and precise identification of pathology in diabetes pregnancy may facilitate important obstetric decisions regarding initiation of insulin therapy and timing of delivery. This is highly important in order to ensure vaginal birth of a healthy, normal size baby at term.

   Compensation This project is covered in the Patient Compensation Association.

ELIGIBILITY:
Inclusion Criteria:

* Age >18 years
* Singleton pregnancy

Exclusion Criteria:

* Fetal malformation or abnormal karyotype
* Maternal height from spine to chest > 43 cm (for technical reasons)
* Sever claustrophobia or any other contradictions to MRI
* Women who do not read or understand Danish

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — Only pregnant women are eligibile
Study Population: Women with pregestational diabetes or uncomplicated pregnancies who meet the above-mentioned inclusion criteria attending their first trimester ultrasound scan at the department of Obstetrics and Gynecology, Aalborg University Hospital.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2020-11-01 (Actual); Primary Completion 2023-06-30 (Estimated); Study Completion 2023-10-31 (Estimated)

PRIMARY OUTCOMES:
Abnormal birth weight | At birth
  Birth weight below or above normal index for gestational age (-22% - +22%)
Preterm delivery | At birth
  Delivery before gestational age 37+0
Cesarean sections | At birth
  Any elective or acute cesarean section
Preeclampsia | 30 weeks before birth or 5 weeks after birth
  Any degree of preeclamsia / eclampsia og HELLP
Placental pathology | Within 1 year after birth
  Any abnormal placenta pathology

CONTACTS AND LOCATIONS:
Overall Officials: Sidsel L Rathcke, MD, Principal Investigator — Aalborg University Hospital
Locations (1):
- Aalborg University Hospital, Department of Obstetrics and Gynecology, Aalborg, Denmark

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Jensen DM, Damm P, Moelsted-Pedersen L, Ovesen P, Westergaard JG, Moeller M, Beck-Nielsen H. Outcomes in type 1 diabetic pregnancies: a nationwide, population-based study. Diabetes Care. 2004 Dec;27(12):2819-23. doi: 10.2337/diacare.27.12.2819. PMID 15562191
- [Background] Gortazar L, Goday A, Flores-Le Roux JA, Sarsanedas E, Paya A, Mane L, Pedro-Botet J, Benaiges D. Trends in prevalence of pre-existing diabetes and perinatal outcomes: a large, population-based study in Catalonia, Spain, 2006-2015. BMJ Open Diabetes Res Care. 2020 Oct;8(1):e001254. doi: 10.1136/bmjdrc-2020-001254. PMID 33106331
- [Background] Lawrence JM, Contreras R, Chen W, Sacks DA. Trends in the prevalence of preexisting diabetes and gestational diabetes mellitus among a racially/ethnically diverse population of pregnant women, 1999-2005. Diabetes Care. 2008 May;31(5):899-904. doi: 10.2337/dc07-2345. Epub 2008 Jan 25. PMID 18223030
- [Background] Persson M, Norman M, Hanson U. Obstetric and perinatal outcomes in type 1 diabetic pregnancies: A large, population-based study. Diabetes Care. 2009 Nov;32(11):2005-9. doi: 10.2337/dc09-0656. Epub 2009 Aug 12. PMID 19675195
- [Background] Yu L, Zeng XL, Cheng ML, Yang GZ, Wang B, Xiao ZW, Luo X, Zhang BF, Xiao DW, Zhang S, Liu HJ, Hu YX, Lei HK, Li QF, Wang ZR. Quantitative assessment of the effect of pre-gestational diabetes and risk of adverse maternal, perinatal and neonatal outcomes. Oncotarget. 2017 May 11;8(37):61048-61056. doi: 10.18632/oncotarget.17824. eCollection 2017 Sep 22. PMID 28977845
- [Background] Evers IM, Nikkels PG, Sikkema JM, Visser GH. Placental pathology in women with type 1 diabetes and in a control group with normal and large-for-gestational-age infants. Placenta. 2003 Sep-Oct;24(8-9):819-25. doi: 10.1016/s0143-4004(03)00128-0. PMID 13129678
- [Background] Evers IM, de Valk HW, Mol BW, ter Braak EW, Visser GH. Macrosomia despite good glycaemic control in Type I diabetic pregnancy; results of a nationwide study in The Netherlands. Diabetologia. 2002 Nov;45(11):1484-9. doi: 10.1007/s00125-002-0958-7. Epub 2002 Sep 25. PMID 12436330
- [Background] Laurini RN, Visser GH, van Ballegooie E, Schoots CJ. Morphological findings in placentae of insulin-dependent diabetic patients treated with continuous subcutaneous insulin infusion (CSII). Placenta. 1987 Mar-Apr;8(2):153-65. doi: 10.1016/0143-4004(87)90018-x. PMID 3615374
- [Background] Jirkovska M, Kucera T, Dvorakova V, Jadrnicek M, Moravcova M, Zizka Z, Krejci V. Impact of maternal diabetes type 1 on proliferative potential, differentiation and apoptotic activity in villous capillaries of term placenta. Placenta. 2016 Apr;40:1-7. doi: 10.1016/j.placenta.2016.02.003. Epub 2016 Feb 9. PMID 27016776
- [Background] Mayhew TM. Enhanced fetoplacental angiogenesis in pre-gestational diabetes mellitus: the extra growth is exclusively longitudinal and not accompanied by microvascular remodelling. Diabetologia. 2002 Oct;45(10):1434-9. doi: 10.1007/s00125-002-0927-1. Epub 2002 Sep 5. PMID 12378385
- [Background] Mayhew TM, Sorensen FB, Klebe JG, Jackson MR. Growth and maturation of villi in placentae from well-controlled diabetic women. Placenta. 1994 Jan;15(1):57-65. doi: 10.1016/s0143-4004(05)80236-x. PMID 8208670
- [Background] Kinsley B. Achieving better outcomes in pregnancies complicated by type 1 and type 2 diabetes mellitus. Clin Ther. 2007;29 Suppl D:S153-60. doi: 10.1016/j.clinthera.2007.12.015. PMID 18191067
- [Background] Baschat AA. Fetal responses to placental insufficiency: an update. BJOG. 2004 Oct;111(10):1031-41. doi: 10.1111/j.1471-0528.2004.00273.x. No abstract available. PMID 15383103
- [Background] Salvesen DR, Higueras MT, Mansur CA, Freeman J, Brudenell JM, Nicolaides KH. Placental and fetal Doppler velocimetry in pregnancies complicated by maternal diabetes mellitus. Am J Obstet Gynecol. 1993 Feb;168(2):645-52. doi: 10.1016/0002-9378(93)90512-h. PMID 8438946
- [Background] Staff AC, Redman CW, Williams D, Leeson P, Moe K, Thilaganathan B, Magnus P, Steegers EA, Tsigas EZ, Ness RB, Myatt L, Poston L, Roberts JM; Global Pregnancy Collaboration (CoLab). Pregnancy and Long-Term Maternal Cardiovascular Health: Progress Through Harmonization of Research Cohorts and Biobanks. Hypertension. 2016 Feb;67(2):251-60. doi: 10.1161/HYPERTENSIONAHA.115.06357. Epub 2015 Dec 14. No abstract available. PMID 26667417
- [Background] Shah BR, Retnakaran R, Booth GL. Increased risk of cardiovascular disease in young women following gestational diabetes mellitus. Diabetes Care. 2008 Aug;31(8):1668-9. doi: 10.2337/dc08-0706. Epub 2008 May 16. PMID 18487472
- [Background] Gunderson EP, Chiang V, Pletcher MJ, Jacobs DR, Quesenberry CP, Sidney S, Lewis CE. History of gestational diabetes mellitus and future risk of atherosclerosis in mid-life: the Coronary Artery Risk Development in Young Adults study. J Am Heart Assoc. 2014 Mar 12;3(2):e000490. doi: 10.1161/JAHA.113.000490. PMID 24622610
- [Background] Vonck S, Staelens AS, Bollen I, Broekx L, Gyselaers W. Why non-invasive maternal hemodynamics assessment is clinically relevant in early pregnancy: a literature review. BMC Pregnancy Childbirth. 2016 Oct 12;16(1):302. doi: 10.1186/s12884-016-1091-9. PMID 27729024
- [Background] Gyselaers W, Thilaganathan B. Preeclampsia: a gestational cardiorenal syndrome. J Physiol. 2019 Sep;597(18):4695-4714. doi: 10.1113/JP274893. Epub 2019 Aug 14. PMID 31343740
- [Background] Rolnik DL, Wright D, Poon LC, O'Gorman N, Syngelaki A, de Paco Matallana C, Akolekar R, Cicero S, Janga D, Singh M, Molina FS, Persico N, Jani JC, Plasencia W, Papaioannou G, Tenenbaum-Gavish K, Meiri H, Gizurarson S, Maclagan K, Nicolaides KH. Aspirin versus Placebo in Pregnancies at High Risk for Preterm Preeclampsia. N Engl J Med. 2017 Aug 17;377(7):613-622. doi: 10.1056/NEJMoa1704559. Epub 2017 Jun 28. PMID 28657417
- [Background] Lorenz CH, Walker ES, Morgan VL, Klein SS, Graham TP Jr. Normal human right and left ventricular mass, systolic function, and gender differences by cine magnetic resonance imaging. J Cardiovasc Magn Reson. 1999;1(1):7-21. doi: 10.3109/10976649909080829. PMID 11550343
- [Background] Seraphim A, Knott KD, Augusto J, Bhuva AN, Manisty C, Moon JC. Quantitative cardiac MRI. J Magn Reson Imaging. 2020 Mar;51(3):693-711. doi: 10.1002/jmri.26789. Epub 2019 May 20. PMID 31111616
- [Background] Hammoud NM, Visser GH, Peters SA, Graatsma EM, Pistorius L, de Valk HW. Fetal growth profiles of macrosomic and non-macrosomic infants of women with pregestational or gestational diabetes. Ultrasound Obstet Gynecol. 2013 Apr;41(4):390-7. doi: 10.1002/uog.11221. Epub 2013 Mar 11. PMID 22744817
- [Background] Hadlock FP, Harrist RB, Sharman RS, Deter RL, Park SK. Estimation of fetal weight with the use of head, body, and femur measurements--a prospective study. Am J Obstet Gynecol. 1985 Feb 1;151(3):333-7. doi: 10.1016/0002-9378(85)90298-4. PMID 3881966
- [Background] Siauve N, Chalouhi GE, Deloison B, Alison M, Clement O, Ville Y, Salomon LJ. Functional imaging of the human placenta with magnetic resonance. Am J Obstet Gynecol. 2015 Oct;213(4 Suppl):S103-14. doi: 10.1016/j.ajog.2015.06.045. PMID 26428488
- [Background] Moore RJ, Issa B, Tokarczuk P, Duncan KR, Boulby P, Baker PN, Bowtell RW, Worthington BS, Johnson IR, Gowland PA. In vivo intravoxel incoherent motion measurements in the human placenta using echo-planar imaging at 0.5 T. Magn Reson Med. 2000 Feb;43(2):295-302. doi: 10.1002/(sici)1522-2594(200002)43:23.0.co;2-2. PMID 10680695
- [Background] Derwig I, Lythgoe DJ, Barker GJ, Poon L, Gowland P, Yeung R, Zelaya F, Nicolaides K. Association of placental perfusion, as assessed by magnetic resonance imaging and uterine artery Doppler ultrasound, and its relationship to pregnancy outcome. Placenta. 2013 Oct;34(10):885-91. doi: 10.1016/j.placenta.2013.07.006. Epub 2013 Aug 9. PMID 23937958
- [Background] Chavhan GB, Babyn PS, Thomas B, Shroff MM, Haacke EM. Principles, techniques, and applications of T2*-based MR imaging and its special applications. Radiographics. 2009 Sep-Oct;29(5):1433-49. doi: 10.1148/rg.295095034. PMID 19755604
- [Background] Avni R, Neeman M, Garbow JR. Functional MRI of the placenta--From rodents to humans. Placenta. 2015 Jun;36(6):615-22. doi: 10.1016/j.placenta.2015.04.003. Epub 2015 Apr 17. PMID 25916594
- [Background] Khong TY, Mooney EE, Ariel I, Balmus NC, Boyd TK, Brundler MA, Derricott H, Evans MJ, Faye-Petersen OM, Gillan JE, Heazell AE, Heller DS, Jacques SM, Keating S, Kelehan P, Maes A, McKay EM, Morgan TK, Nikkels PG, Parks WT, Redline RW, Scheimberg I, Schoots MH, Sebire NJ, Timmer A, Turowski G, van der Voorn JP, van Lijnschoten I, Gordijn SJ. Sampling and Definitions of Placental Lesions: Amsterdam Placental Workshop Group Consensus Statement. Arch Pathol Lab Med. 2016 Jul;140(7):698-713. doi: 10.5858/arpa.2015-0225-CC. Epub 2016 May 25. PMID 27223167
- [Background] Tee LM, Kan EY, Cheung JC, Leung WC. Magnetic resonance imaging of the fetal brain. Hong Kong Med J. 2016 Jun;22(3):270-8. doi: 10.12809/hkmj154678. Epub 2016 Apr 22. PMID 27101791
- [Background] Clements H, Duncan KR, Fielding K, Gowland PA, Johnson IR, Baker PN. Infants exposed to MRI in utero have a normal paediatric assessment at 9 months of age. Br J Radiol. 2000 Feb;73(866):190-4. doi: 10.1259/bjr.73.866.10884733.
- [Background] Baker PN, Johnson IR, Harvey PR, Gowland PA, Mansfield P. A three-year follow-up of children imaged in utero with echo-planar magnetic resonance. Am J Obstet Gynecol. 1994 Jan;170(1 Pt 1):32-3. doi: 10.1016/s0002-9378(94)70379-5. PMID 8296840
- [Background] Price DL, De Wilde JP, Papadaki AM, Curran JS, Kitney RI. Investigation of acoustic noise on 15 MRI scanners from 0.2 T to 3 T. J Magn Reson Imaging. 2001 Feb;13(2):288-93. doi: 10.1002/1522-2586(200102)13:23.0.co;2-p. PMID 11169836
- [Background] Glover P, Hykin J, Gowland P, Wright J, Johnson I, Mansfield P. An assessment of the intrauterine sound intensity level during obstetric echo-planar magnetic resonance imaging. Br J Radiol. 1995 Oct;68(814):1090-4. doi: 10.1259/0007-1285-68-814-1090. PMID 7496710
- [Background] Strizek B, Jani JC, Mucyo E, De Keyzer F, Pauwels I, Ziane S, Mansbach AL, Deltenre P, Cos T, Cannie MM. Safety of MR Imaging at 1.5 T in Fetuses: A Retrospective Case-Control Study of Birth Weights and the Effects of Acoustic Noise. Radiology. 2015 May;275(2):530-7. doi: 10.1148/radiol.14141382. Epub 2015 Jan 7. PMID 25575119
- [Background] Bouyssi-Kobar M, du Plessis AJ, Robertson RL, Limperopoulos C. Fetal magnetic resonance imaging: exposure times and functional outcomes at preschool age. Pediatr Radiol. 2015 Nov;45(12):1823-30. doi: 10.1007/s00247-015-3408-7. Epub 2015 Jul 9. PMID 26155983
- [Background] International Commission on Non-Ionizing Radiation Protection (ICNIRP). Medical magnetic resonance (MR) procedures: protection of patients. Health Phys. 2004 Aug;87(2):197-216. doi: 10.1097/00004032-200408000-00008. No abstract available. PMID 15257220
- [Background] Kangarlu A, Burgess RE, Zhu H, Nakayama T, Hamlin RL, Abduljalil AM, Robitaille PM. Cognitive, cardiac, and physiological safety studies in ultra high field magnetic resonance imaging. Magn Reson Imaging. 1999 Dec;17(10):1407-16. doi: 10.1016/s0730-725x(99)00086-7. PMID 10609989
- [Background] Poutamo J, Partanen K, Vanninen R, Vainio P, Kirkinen P. MRI does not change fetal cardiotocographic parameters. Prenat Diagn. 1998 Nov;18(11):1149-54. doi: 10.1002/(sici)1097-0223(199811)18:113.0.co;2-k. PMID 9854723
- [Background] Michel SC, Rake A, Keller TM, Huch R, Konig V, Seifert B, Marincek B, Kubik-Huch RA. Original report. Fetal cardiographic monitoring during 1.5-T MR imaging. AJR Am J Roentgenol. 2003 Apr;180(4):1159-64. doi: 10.2214/ajr.180.4.1801159. PMID 12646475
- [Background] International Commission on Non-Ionizing Radiation Protection (ICNIRP). Guidelines for limiting exposure to time-varying electric and magnetic fields (1 Hz to 100 kHz). Health Phys. 2010 Dec;99(6):818-36. doi: 10.1097/HP.0b013e3181f06c86. No abstract available. PMID 21068601
- [Background] International Commission on Non-Ionizing Radiation Protection (ICNIRP). Amendment to the ICNIRP "Statement on medical magnetic resonance (MR) procedures: protection of patients". Health Phys. 2009 Sep;97(3):259-61. doi: 10.1097/HP.0b013e3181aff9eb. No abstract available. PMID 19667810
- [Background] Hand JW, Li Y, Thomas EL, Rutherford MA, Hajnal JV. Prediction of specific absorption rate in mother and fetus associated with MRI examinations during pregnancy. Magn Reson Med. 2006 Apr;55(4):883-93. doi: 10.1002/mrm.20824. PMID 16508913
- [Background] Abramowicz JS, Barnett SB, Duck FA, Edmonds PD, Hynynen KH, Ziskin MC. Fetal thermal effects of diagnostic ultrasound. J Ultrasound Med. 2008 Apr;27(4):541-59; quiz 560-3. doi: 10.7863/jum.2008.27.4.541. PMID 18359908
- [Background] Sheiner E, Freeman J, Abramowicz JS. Acoustic output as measured by mechanical and thermal indices during routine obstetric ultrasound examinations. J Ultrasound Med. 2005 Dec;24(12):1665-70. doi: 10.7863/jum.2005.24.12.1665. PMID 16301723
- See also: DSOG. Patoanatomisk Undersøgelse af Placenta [Internet]. 2016. Available from: http://gynobsguideline.dk/sandbjerg/Patoanatomi placenta.pdf — http://gynobsguideline.dk/sandbjerg/Patoanatomi%20placenta.pdf